CLINICAL TRIAL: NCT04504279
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, 16-Week Trial to Evaluate the Efficacy and Safety of FB-401 in Children, Adolescent and Adult Subjects (Ages 2 Years and Older) With Mild to Moderate Atopic Dermatitis
Brief Title: Evaluation of FB-401 in Children, Adolescents and Adults (2 Years and Older) With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forte Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB401-01
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; microbiome; probiotic; commensal Gram-negative bacteria; transdermal water loss; allergic diseases; dermatitis; eczema; skin diseases; skin diseases, eczematous; immune system diseases
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Skin Diseases, Eczematous; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FB-401 (Experimental): FB-401 applied topically for 16 weeks.
  Interventions: Biological: FB-401
- Placebo (Placebo Comparator): Placebo applied topically for 16 weeks.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: FB-401 — Topical application
  Arms: FB-401
Biological: Placebo — Vehicle
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential improvement in atopic dermatitis signs and symptoms following the application of FB-401 in patients 2 years or older with mild to moderate atopic dermatitis. FB-401 will be applied topically for 16 weeks and progress will be assessed by assessment of the skin and patient reports.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 2 years of age
* Clinical diagnosis of atopic dermatitis as defined by Hanifin and Rajka criteria that has been present for ≥ 3 months before the screening visit
* Investigator Global Assessment (IGA) score of 2 (mild) or 3 (moderate) at Screening and Baseline/Day 1 using the validated IGA scale for atopic dermatitis
* EASI score ≥ 5 at the screening and the Baseline visit
* 5% to 30% (inclusive) body surface area of atopic dermatitis involvement at the screening and the baseline visit

Exclusion Criteria:

* Previous treatment within 4 weeks prior to the baseline visit with any of the following:
* Immunosuppressive or immunomodulating systemic drugs such as systemic (intravenous, oral, intra-articular or intramuscular) corticosteroids, azathioprine, methotrexate, cyclosporine
* Phototherapy or photo chemotherapy for atopic dermatitis
* Previous treatment within 1 week prior to the baseline visit with any of the following:
* Topical corticosteroids (does not include inhaled, intranasal or ophthalmic) or topical calcineurin inhibitors
* Topical phosphodiesterase type 4 (PDE4) inhibitor
* Use of emollients other than provided for the study
* Bleach baths
* Within 8 weeks or 5 half-lives (if known), whichever is longer, prior to the baseline visit with Janus kinase inhibitors or other investigational drug
* Within16 weeks or 5 half-lives, whichever is longer, prior to the baseline visit with dupilumab or other biologic agent to treat atopic dermatitis
* Within 1 year prior to the baseline visit with any live bacterial therapy
* Pregnant (or planning to become pregnant during the period of the study) or lactating females

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
EASI 50 | 16 weeks
  The proportion of subjects with 50% improvement in Eczema Area and Severity Index (EASI) score from baseline at Week 16

SECONDARY OUTCOMES:
Includes percent change in EASI | 16 weeks
  Percent change in EASI score is measured from baseline to Week 16

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - DS Research, Clarksville, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - DS Research, Louisville, Kentucky
  - Lawrence J. Green MD LLC, Rockville, Maryland
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - Cyn3rgy Research, Gresham, Oregon
  - KGL Skin Study Center LLC, Newtown Square, Pennsylvania
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myles IA, Earland NJ, Anderson ED, Moore IN, Kieh MD, Williams KW, Saleem A, Fontecilla NM, Welch PA, Darnell DA, Barnhart LA, Sun AA, Uzel G, Datta SK. First-in-human topical microbiome transplantation with Roseomonas mucosa for atopic dermatitis. JCI Insight. 2018 May 3;3(9):e120608. doi: 10.1172/jci.insight.120608. PMID 29720571